CLINICAL TRIAL: NCT03772405
Title: Cross Over Study to Assess the Effect of the Nasal Gel "Nascum®-Plus" on Allergic Symptoms and Inflammatory Cells and Cytokines During and After Allergen Challenge in the Fraunhofer Allergen Challenge Chamber (ACC)
Brief Title: Effect of the Nasal Gel "Nascum®-Plus" on Allergic Symptoms
Acronym: NAPO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fraunhofer-Institute of Toxicology and Experimental Medicine (Other)
Collaborators: M et P Pharma AG (Unknown)
Responsible Party: Principal Investigator, Philipp Badorrek, Head of Department, Principle Investigator, Fraunhofer-Institute of Toxicology and Experimental Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-05 NAPO
Record Dates: First submitted 2018-12-10; First posted 2018-12-11 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Rhinitis, Allergic, Seasonal
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nascum Plus and ACC (Experimental): In a cross-over design, patients are exposed to pollen in the ACC twice for 4 hours each 3 weeks apart. Subjects will receive treatment with Nascum Plus either 5 minutes before the first or the second 4 hour pollen challenge.
  Interventions: Drug: Nascum Plus; Other: ACC

INTERVENTIONS:
Drug: Nascum Plus — nasal application of nascum plus
Other: ACC — 4 hours challenge to grass pollen in the allergen challenge chamber (ACC)

SUMMARY:
The aim of this study is to assess if a physical barrier, created by the nasal gel Nascum®- Plus, is able to prevent or minimize the induction of nasal symptoms during allergen challenge in the Fraunhofer Allergen Challenge Chamber (ACC). Furthermore, the effect on soluble and cellular inflammatory markers induced by the allergic reaction will be assessed. Nascum®-Plus contains no active pharmaceutical ingredient, only monographed pharmaceutical excipients.

ELIGIBILITY:
Inclusion Criteria:

* 1. Able and willing to give written informed consent.
* 2. Male and female subjects, aged 18-65 years. Women will be considered for inclusion if they are: Not pregnant, as confirmed by pregnancy test (see flow chart), and not nursing. Of non-child bearing potential (i.e. physiologically incapable of becoming pregnant, including any female who is pre-menarchial or post-menopausal, with documented proof of hysterectomy or tubal ligation, or meets clinical criteria for menopause and has been amenorrhoeic for more than 1 year prior to the screening visit).

Of childbearing potential and using a highly effective method of contraception during the entire study (vasectomised partner, sexual abstinence - the lifestyle of the female should be such that there is complete abstinence from intercourse from two weeks prior to the first dose of study medication until at least 72 hours after treatment -, implants, injectables, combined oral contraceptives, hormonal IUDs or double-barrier methods, i.e. any double combination of IUD, condom with spermicidal gel, diaphragm, sponge, and cervical cap).

* 3. Body mass index between 18 and 32 kg/m²
* 4. History of seasonal allergic rhinitis to grass pollen
* 5. Positive skin prick test for Dactylis glomerata pollen at screening or within 12 months prior to the screening visit.
* 6. Normal lung function Forced Expiratory Volume in one second (FEV1) ≥ 80 % pred and FEV1/Forced Vital Capacity (FVC) >70% at screening
* 7. Adequate level of rhinitis symptoms in a grass pollen challenge, defined as a Total Nasal Symptom Score (TNSS) of at least 6 (of 12) within the 2-hour grass pollen challenge at performed at the Screening ACC visit (V2).
* 8. TNSS of 3 prior to entering the pollen chamber at screening.
* 9. Non-smokers or ex-smokers since at least 6 months with a history of less than 10 pack years

Exclusion Criteria:

* 1. Any clinically relevant abnormal findings in physical examination, clinical chemistry, hematology, urine analysis, vital signs, lung function or Electrocardiogram (ECG) at screening visit , which, in the opinion of the investigator, may either put the subject at risk because of participation in the study or may influence the results of the study, or the subject's ability to participate in the study
* 2. Past or present disease, which as judged by the investigator, may affect the outcome of this study. These diseases include, but are not limited to, cardiovascular disease, malignancy, hepatic disease, renal disease, hematological disease, neurological disease, endocrine disease or pulmonary disease (including but not confined to chronic bronchitis, emphysema, tuberculosis, bronchiectasis or cystic fibrosis).
* 3. History of an acute infection four weeks prior to the informed consent visit
* 4. Specific Immunotherapy (SIT) within 2 years prior to the study
* 5. Rhinitis of other cause, chronic sinusitis or rhinitis or sinusitis in the last 14 days before entering the study
* 6. Asthma requiring more than inhaled short-acting beta-2 agonists.
* 7. Conditions or factors, which would make the subject unlikely to be able to stay in the Fraunhofer ACC for 4 hours.
* 8. Any contraindication for adrenalin use (e.g. use of local and systemic beta-blockers, angiotensin-converting-enzyme (ACE) inhibitors
* 9. Treatment with antipsychotic medications with antihistaminic effect (e.g. chlorpromazine, levomepromazine, clozapine, olanzapine, tioridazine)
* 10. Use of any medications according to section 8.2 in the period indicated before allergen challenge
* 11. Participation in another clinical trial 30 days prior to enrollment.
* 12. History of drug or alcohol abuse
* 13. Risk of non-compliance with study procedures
* 14. Suspected inability to understand the protocol requirements, instructions and study-related restrictions, the nature, scope, and possible consequences of the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2018-12-12 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
Total Nasal Symptom Score (TNSS) | pre start of challenge and every 20 minutes during 4 hours challenge
  Change of TNSS assessed during grass pollen challenge in ACC

CONTACTS AND LOCATIONS:
Overall Officials: Philipp Badorrek, MD, Principal Investigator — The Fraunhofer-Gesellschaft
Locations (1):
- Fraunhofer ITEM, Hanover, Lower Saxony, Germany